CLINICAL TRIAL: NCT04610957
Title: Effect of Adding Isoflavonoids to Clomiphene Citrate for Ovulation Induction in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FAlbasri (Other Government)
Responsible Party: Sponsor-Investigator, FAlbasri, Resident of Obstetrics and Gynecology, Alkhoms Hospital, Misurata University, Libya, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5111
Record Dates: First submitted 2020-10-01; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Ovulation Induction; Polycystic Ovary Syndrome
Keywords: Human chorionic gonadotropin; clomiphene Citrate; Isoflavonoids; polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The 1st group (Experimental): included eighty (80) women receiving Clomiphene citrate (CC) in the form of (Clomid 50 mg tablet, Sanofi Aventis, France) at dose (100 mg/day in two divided doses, starting from day 3 to day 7 of the cycle), plus Phytoestrogens (Isoflavonoids) in the form of (RosaFem 800 mg tablet, DeluxLab, Egypt) at dose (1600 mg/day in two divided doses (each dose one tablet), starting from day 3 to day 12 of the cycle
  Interventions: Drug: Rosafem (FEMININE FORMULA)
- The 2nd group (Experimental): included eighty (80) women receiving Clomiphene citrate only, at dose (100 mg/day, starting from day 3 to day 7 of the cycle).
  Interventions: Drug: Rosafem (FEMININE FORMULA)

INTERVENTIONS:
Drug: Rosafem (FEMININE FORMULA) — Rosafem is the only phytoestrogen product with the convenient dose which provides significant improvement of menopausal related symptoms premenstrual syndrome symptoms

SUMMARY:
This prospective, randomized clinical trial double blinded study, has been carried on 160 infertile patients seeking pregnancy in Gynecology and Obstetrics Department, Zagazig University Hospitals during the period from January 2019 to November 2019, the participants' randomizations were done and patients divided into two groups; group I: included 80 women receiving Clomiphene citrate (CC) plus Isoflavonoids. Group 2: included 80 women receiving Clomiphene citrate only

DETAILED DESCRIPTION:
Phytoestrogens continue to be of increasing interest because of their possible influence on the physiology of the reproductive tract.

The aim of Prospective randomized clinical trial study is to evaluate effect of adding isoflavonoids to clomiphene citrate during ovulation induction in women with PCOS on the endometrial thickness which has an impact on pregnancy rate.

This study included 160 infertile women seeking pregnancy and they were divided into two groups. Clomiphene is given orally at dose, one tablet twice per day (tablet 50 mg), from day 3 to day 7 for all patients (group I and group II),while phytoestrogens are given at dose, two tablets two times per day (tablet 800mg), from day 3 to day 12 only for group I, followed by HCG injection on attaining mature follicle(s) by trans-vaginal US scan with diameter ≥ 18 mm.

ELIGIBILITY:
Inclusion Criteria:

• Patient aged 18- 35 years old with primary or secondary infertility

Exclusion Criteria:

* Patient aged 18- 35 years old with primary or secondary infertility
* Patient whose husband has a male factor of infertility.
* Hepatic, renal, diabetic, thyroid or cardiovascular disorders.
* Organic pelvic disease (uterine fibroids or ovarian cysts).
* Abnormality detected by HSG as blocked tubes

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | up to 24 weeks
  defined as the presence of gestational sac containing fetal hearts on ultrasound scan

SECONDARY OUTCOMES:
Endometrial thickness, | up to 24 weeks
  endometrial thickness is used to monitor infertility treatment
ovulation rate | up to 24 weeks
  Ovulation rate was taken as the gold standard for assessment of ovulation induction result

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No